CLINICAL TRIAL: NCT05095441
Title: A Phase 1 Open-Label Study of Genetically Engineered Oncolytic HSV-1 (C5252) Expressing IL-12 and Anti-PD-1 Antibody in Patients With Recurrent or Progressive Glioblastoma
Brief Title: A Clinical Study of Intratumoral MVR-C5252 (C5252) in Patients With Recurrent or Progressive Glioblastoma
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: ImmVira Pharma Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MVR-C5252-001
Record Dates: First submitted 2021-09-15; First posted 2021-10-27 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Solid Tumor; Glioblastoma; Glioblastoma Multiforme; Glioblastoma Multiforme of Brain
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1: Dose Escalation (Experimental): C5252 single agent dose escalation in participants with glioblastoma
  Interventions: Biological: C5252
- Part 2: Dose Expansion (Experimental): Recommended dose of C5252 as determined in Part 1 Dose Escalation in participants with glioblastoma
  Interventions: Biological: C5252

INTERVENTIONS:
Biological: C5252 — A single dose of C5252 will be administered up to 2mL as intratumoral injection on Day 1.

SUMMARY:
This is a Phase 1 open label, first in human study of C5252 monotherapy designed to determine the safety and tolerability of a single intratumoral (IT) injection of C5252 in patients with recurrent or progressive glioblastoma (GBM).

DETAILED DESCRIPTION:
This is a Phase 1 open label, first in human study of C5252 monotherapy designed to determine the safety and tolerability of a single IT injection of C5252 in patients with recurrent or progressive GBM. The Part 1 portion of the study is a 3+3 design to evaluate escalating doses of C5252. Total enrollment will depend on the toxicities and/or activity observed, with approximately 36 evaluable participants enrolled. Once the recommended dose (RD) is identified from Part 1, Part 2 Dose Expansion will enroll up to 15 additional participants to further assess the safety, tolerability, and preliminary efficacy of a single IT injection of C5252 monotherapy.

ELIGIBILITY:
Key Inclusion Criteria:

1. Signed and dated approved informed consent form (ICF) before any protocol-directed screening procedures are performed.
2. Participants must have histopathologically confirmed recurrent supratentorial glioblastoma.
3. Participants must have progressed after at least 1 line but no more than 2 lines of therapy.
4. Evidence of progression by RANO criteria based on MRI scan.
5. Residual lesion must be ≥ 1.0 cm and < 5.5 cm contrast-enhancing in diameter as determined by MRI.
6. Age ≥ 18 years.
7. Karnofsky Performance Score (KPS) ≥ 70.
8. Life expectancy > 12 weeks.
9. Participants must have normal organ and marrow function.
10. Participants must commit to the use of a reliable method of birth control.
11. Resolution of all AEs due to previous therapies to ≤ Grade 1 or baseline.
12. Capable of understanding and complying with protocol requirements.

Key Exclusion Criteria:

1. Inability to undergo MRI examination for any reason.
2. A contrast-enhancing brain tumor that does not meet protocol criteria.
3. Prior history of encephalitis, multiple sclerosis, or other CNS infection.
4. Clinical diagnosis of Li-Fraumeni Syndrome or with a known germ line deficit in the retinoblastoma gene or its related pathways.
5. Required steroid increase within 2 weeks prior to date of C5252 administration.
6. Systemic therapy with immunosuppressive agents within 28 days prior to date of C5252 administration.
7. Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or any other medical condition that precludes surgery. Also, psychiatric illness/social situations that would limit compliance with study requirements.
8. Bleeding diathesis, or requirement for anticoagulants, or antiplatelet agents, including NSAIDs that cannot be stopped for surgery or biopsy.
9. Current diagnosis of other cancer except in situ cervical cancer, basal or squamous cell carcinoma of the skin.
10. Requires continued concurrent therapy with any drug active against HSV (acyclovir, valaciclovir, penciclovir, famciclovir, ganciclovir, foscarnet, cidofovir).
11. Pregnant or lactating.
12. Prior organ transplantation.
13. Active hepatitis B virus, hepatitis C virus, or a positive serological test at Screening.
14. Active oral herpes lesion at Screening.
15. Congestive heart failure (> New York Heart Association Class II), active coronary artery disease, unevaluated new onset angina within 3 months or unstable angina (angina symptoms at rest), or clinically significant cardiac arrhythmias.
16. History of allergic reactions attributed to compounds of similar biological composition to HSV-1, IL-12, or anti-PD-1 monoclonal antibody.
17. Active infection with SARS-CoV-2 virus.
18. Other systemic conditions or organ abnormalities that, in the opinion of the Investigator, may interfere with the conduct and/or interpretation of the current study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2023-03-15 (Estimated); Primary Completion 2023-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate the safety and tolerability of C5252 | Up to 28 days from C5252 injection
  Number of participants in dose escalating cohorts with dose limiting toxicities (DLTs), treatment-emergent adverse events (TEAEs), and/or changes in clinical laboratory abnormalities.
Characterize Dose Limiting Toxicities | Up to 28 days from C5252 injection
  Incidence of DLTs
Identify the maximum tolerated dose (MTD) and/or the RD of C5252 | Up to 28 days from C5252 injection
  Incidence of DLTs

SECONDARY OUTCOMES:
Evaluate the PK of C5252 | Up to 2 years from C5252 injection
  Measure anti-PD-1 antibody concentration in blood using Anti-PD-1 antibody ELISA test and IL-12 concentration in blood using IL-12p70 ELISA test.
Evaluate the viral shedding of C5252 | Up to 2 years from C5252 injection
  Measure viral shedding of C5252 after intratumoral injection in saliva, nasopharyngeal mucus, and urine using qPCR (quantitative polymerase chain reaction) test.
Overall response rate (ORR) | Up to 2 years from C5252 injection
  ORR is defined as the proportion of participants who have had a partial response (PR), or complete response (CR) to intervention, based on Investigator Assessment for Neuro-oncology (RANO).
Progression-free survival (PFS) | Up to 2 years from C5252 injection
  PFS is defined as the time from Day 1 to the first documentation of progressive disease (PD) or death from any cause, whichever occurs first per RANO.
Overall Survival (OS) | Up to 2 years from C5252 injection
  OS is defined as the time from enrollment to death from any cause.

OTHER OUTCOMES:
Evaluate blood cytokines | Up to 28 days from C5252 injection
  Measure blood cytokines using MSD V-Plex Electrochemiluminescence Immunoassay test.
Evaluate lymphocyte profiling | Up to 28 days from C5252 injection
  Conduct lymphocyte profiling using PBMC Flow cytometry test.

CONTACTS AND LOCATIONS:
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No